CLINICAL TRIAL: NCT01164644
Title: The Utility of Peri-operative Arnica Montana for Reduction of Ecchymosis in Rhinoplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2010-0065
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Ecchymosis
Keywords: ecchymosis; bruising; rhinoplasty; nose job; arnica; arnica montana
MeSH Terms: conditions — Ecchymosis; Contusions | interventions — Arnicae flos extract; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arnica Montana (Active Comparator): The subject will take twelve pills by mouth three times a day over four days.
  Interventions: Drug: Arnica montana
- Placebo (Placebo Comparator): The subject will take twelve pills by mouth three times a day over four days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arnica montana — Subjects will take twelve pills by mouth three times a day over four days.
  Arms: Arnica Montana
Drug: Placebo — Subjects will take twelve pills by mouth three times a day over four days.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Arnica montana is a homeopathic drug that is made in accordance with the official methods of the Homeopathic Pharmacopoeia of the United States (HPUS) and is commonly used by cosmetic surgeons throughout the world, although there is no study proving its benefit after rhinoplasty surgery. The purpose of the research is to see if Arnica montana will reduce the amount of bruising and the intensity of the bruising after surgery. Photographs of the subject's face will be taken and used to analyze bruising after rhinoplasty surgery in subjects who receive Arnica montana and compare them to photographs of subjects who take a placebo (sugar pill).

DETAILED DESCRIPTION:
Subjects will receive either oral arnica montana or placebo without any identifying labels or markers on the drugs.

During the post-operative period, the patients will be seen back in surgery clinic on post-operative days 3, 7 and 10. During the first two visits, the subject will receive routine post-operative care with no difference from patients not enrolled in the study. This includes routine sets of photographs. The participant will then return for a third post-operative visit lasting under ten minutes only for study photos using the left and right "three-quarters" view. Again, the subject will hold a measurement marker so length measurements can be made, and this marker will be held under the ear to not interfere with the routine cosmetic analysis of the photographs. The digital photographs will be used to analyze the bruising for the study. The ratio was calculated by dividing the number of pixels of bruised area over number of pixels of standard area.

ELIGIBILITY:
Inclusion Criteria: Adult patients who are deemed candidates for rhinoplasty surgery at UW Transformations will be eligible to participate in the study.

-

Exclusion Criteria:

* Patients who are prisoners
* Patients who are pregnant and breast-feeding women
* Patients taking anti-coagulants (such as blood thinners), anti-platelet drugs (such as NSAIDS), or other homeopathic remedies during the peri-operative period
* Patients with a bruising or bleeding disorder
* Patients who take oral corticosteroid therapy
* Patients who suffer from severe liver or kidney disease
* Patients with malignancy, infection, immunodeficiency, metabolic syndrome, infectious or inflammatory gastrointestinal disease
* Patients with oral or contact allergies to Arnica montana or to any other member of the Asteraceae family of plants such as ragweed, chrysanthemums, marigolds, and daisies

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin C Marcus, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients scheduled for rhinoplasty surgery with nasal bone osteotomies by the senior author at an outpatient surgery center were recruited by a clinic nurse practitioner (GJ) during the routine pre-operative history and physical exam visit. Enrollment was opened from July of 2009 through June of 2012.
Pre-assignment Details: 28 subjects were recruited, 22 completed the study. One elected to leave the study prior to surgery, 2 attended only one post-operative visit; 2 did not undergo surgery (loss of health insurance [1] and thrombocytopenia [1]); and 1 subject elected to leave the study for laser treatments for ecchymosis on post-operative day 3
Period: Overall Study
Arm/Group | Arnica Montana | Placebo
Started | 12 | 14
Completed | 9 | 13
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arnica Montana | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.75 (13.06) | 32.71 (13.34) | 33.65 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Assess Extent of Bruising
Description: Primary outcome measure will be to measure the extent of bruising in based on a ratio of pixels on post-operative day number three. Every subject held a card in front of their face with a specific size marker. The square area of this marker was known and used to measure the number of pixels in this marker with Photoshop and compare it to the known area. Next the area of bruising was measured in number of pixels. Therefore for every photograph a standardized ratio of pixels was known because of the marker. The ratio was calculated by dividing the number of pixels of bruised area over number of pixels of standard area.
Time Frame: Post-operative day 3
Measure: Mean (Standard Error); unit: a ratio of pixels
Arm/Group | Arnica Montana | Placebo
Number analyzed (Participants) | 9 | 13
a ratio of pixels | .617 (.091) | .736 (.118)

2. Primary Outcome: Assess Extent of Bruising
Description: Primary outcome measure will be to measure the extent of bruising based on a ratio of pixels on post-operative day number seven. Every subject held a card in front of their face with a specific size marker. The square area of this marker was known and used to measure the number of pixels in this marker with Photoshop and compare it to the known area. Next the area of bruising was measured in number of pixels. Therefore for every photograph a standardized ratio of pixels was known because of the marker.
Time Frame: Post-operative day 7
Measure: Mean (Standard Error); unit: a ratio of pixels
Arm/Group | Arnica Montana | Placebo
Number analyzed (Participants) | 9 | 13
a ratio of pixels | .600 (.082) | .894 (.146)

3. Primary Outcome: Assess Extent of Bruising
Description: Primary outcome measure will be to measure the extent of bruising based on a ratio of pixels on post-operative day number ten. Every subject held a card in front of their face with a specific size marker. The square area of this marker was known and used to measure the number of pixels in this marker with Photoshop and compare it to the known area. Next the area of bruising was measured in number of pixels. Therefore for every photograph a standardized ratio of pixels was known because of the marker.
Time Frame: Post-operative day 10
Measure: Mean (Standard Error); unit: a ratio of pixels
Arm/Group | Arnica Montana | Placebo
Number analyzed (Participants) | 9 | 13
a ratio of pixels | .432 (.125) | .543 (.094)

ADVERSE EVENTS:
Arm/Group | Arnica Montana | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arnica Montana (N=12) | Placebo (N=14)
thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes